CLINICAL TRIAL: NCT00118781
Title: Randomized, Double-Blind, Placebo-Controlled, Multinational Phase 3 Trial Of Iseganan In Prevention Of Ventilator-Associated Pneumonia
Brief Title: Trial of Iseganan in Prevention of Ventilator-Associated Pneumonia
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: IntraBiotics Pharmaceuticals (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 09-002
Record Dates: First submitted 2005-07-01; First posted 2005-07-12 (Estimated); Last update posted 2005-07-19 (Estimated); Status verified 2005-07

CONDITIONS: Pneumonia
Keywords: ventilator-associated pneumonia; VAP; pneumonia; ICU infection
MeSH Terms: conditions — Pneumonia; Pneumonia, Ventilator-Associated

INTERVENTIONS:
Drug: iseganan hydrochloride

SUMMARY:
This is a multinational, double-blind, placebo-controlled trial designed to assess whether iseganan, applied topically to the oral cavity, can prevent ventilator-associated pneumonia among patients who are intubated and mechanically ventilated and survive for up to 14 days.

DETAILED DESCRIPTION:
Patients will be randomized and receive their first dose of Study Drug within 24 hours of oral/nasal intubation and the initiation of mechanical ventilation. The Study Period will begin with the first administration of Study Drug (Study Day 1). Three mL of Study Drug (9 mg iseganan or matching placebo) will be applied to all visible surfaces in the oral cavity and the oral portion of the endotracheal tube (for non-tracheostomy patients) every 4 hours through Study Day 14, or until the diagnosis of microbiologically-confirmed pneumonia (based on central laboratory results) or extubation, whichever occurs first.

All patients will be evaluated for clinically defined pneumonia at least once daily and, if diagnosed, blood specimens will be collected and cultured, and a bronchoscopic alveolar lavage (BAL) specimen (for intubated patients) or a respiratory secretion specimen (for extubated patients) will be obtained PRIOR to initiating or changing any systemic antimicrobial therapy.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age
* Orally/nasally intubated and receiving mechanical ventilation for <24 hours prior to scheduled randomization and administration of the first dose of Study Drug, and in the judgment of the attending physician, expected to remain intubated and mechanically ventilated for at least 48 hours
* Expected to survive for at least 21 days and to remain at the investigational site and not transferred to another institution while intubated during the 21-day study period
* Willing and able to provide written informed consent, or if unconscious or have altered sensorium, have a surrogate provide written informed consent as approved by the institution
* Negative pregnancy test within 7 days prior to randomization if a female of childbearing potential (Negative pregnancy test results [urine or serum] obtained for reason other than the purposes of this study are acceptable.)

Exclusion Criteria:

* Current diagnosis of pneumonia (Patients currently receiving antibiotics for treatment of pneumonia and patients who meet the study definition of clinically defined pneumonia at the time of screening will be excluded.)
* Absolute neutrophil count less than 1000/mm3
* Human immunodeficiency virus infection with a last known CD4 count less than 500/mm3
* Recipient of organ transplantation and receiving immunosuppressive therapy
* Current hematologic malignancy
* Previously documented cystic fibrosis
* Severe cranio-facial trauma or other medical condition expected to require imminent tracheostomy
* Patient, patient's family and/or physician not in favor of aggressive medical management or presence of an advanced directive to withhold life-sustaining treatment
* Moribund state or expected to survive less than 21 days due to an uncorrectable medical condition
* Participation in a clinical trial of any unlicensed drug, biologic or device within 30 days prior to the first dose of study drug
* Concurrent participation in a clinical trial of any unlicensed drug, biologic or device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900
Dates: Start 2003-09; Study Completion 2004-06

PRIMARY OUTCOMES:
The primary objectives of this trial are to evaluate the safety and efficacy of iseganan when administered to intubated patients receiving mechanical ventilation.

SECONDARY OUTCOMES:
The secondary objectives of this trial are to compare patients receiving iseganan to patients receiving placebo on the following: VAP-free survival through Day 21
Days alive and free of parenteral antibiotic use through Day 14
Days alive and free of mechanical ventilation through Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Marin Kollef, MD, Study Chair — Barnes-Jewish Hospital, Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States